CLINICAL TRIAL: NCT03469245
Title: Validation of Fenestrations Positioning by Numerical Simulation in Fenestrated Endovascular Repair of Abdominal Aortic Aneurysms
Brief Title: Validation of Fenestrations Positioning by Numerical Simulation
Acronym: FenSim
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Predisurge Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRBN762017
Record Dates: First submitted 2018-02-19; First posted 2018-03-19 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Endovascular; Fenestrated endovascular repair; numerical simulation
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- abdominal aortic aneurysms treated by fenestrated endovascular: Patients have an abdominal aortic aneurysms treated by fenestrated endovascular anacondaTM of society Vascutek will be included. Predisurge society will perform numerical simulation.
  Interventions: Other: numerical simulation

INTERVENTIONS:
Other: numerical simulation — After patients have been treated by fenestrated endovascular of society Vascutek data will be collected by society Vascutek and send to Predisurge society. They will perform numerical simulation and compare with the method of Vascutek.

SUMMARY:
Fenestrated endovascular repair (FEVAR) is nowadays a recognized option to treat juxtarenal, pararenal or suprarenal abdominal aortic aneurysms in patients at high risk for conventional repair. The technique consists in deploying a custom-made stent-graft (SG) inside the patient aorta. Part of the customization involves cauterizing a hole in SG fabric and reinforcing it with a Nitinol stent ring, thereby creating a fenestration for each corresponding collateral artery. For this reason, preoperative planning is crucial to determine adequate positions of fenestrations, in order to obtain perfect alignment with the collateral arteries of the patient. Inadequate positioning may result in failure to catheterize a collateral artery and subsequent organ damage, increased catheterizing time, increased irradiation dose, endoleaks… The current process of fenestrations positioning for fenestrated anacondaTM SG involves: (i) anatomical measurements on patient preoperative CT-scan by case planners using dedicated sizing software; (ii) designing an initial custom device scheme with its positioned fenestrations, created by engineers with CAD software using the above cited measurements and (iii) validation of fenestrations position by in vitro testing using a SG prototype deployed inside a transparent anatomy model (3D-printed model of patient aorta and collateral arteries). The main limitations of this process are the costs and long SG delivery time.

DETAILED DESCRIPTION:
The current process of fenestrations positioning for fenestrated anacondaTM SG involves: (i) anatomical measurements on patient preoperative CT-scan by case planners using dedicated sizing software; (ii) designing an initial custom device scheme with its positioned fenestrations, created by engineers with CAD software using the above cited measurements and (iii) validation of fenestrations position by in vitro testing using a SG prototype deployed inside a transparent anatomy model (3D-printed model of patient aorta and collateral arteries). The main limitations of this process are the costs and long SG delivery time.

The goal of this study is to compare fenestrations positioning obtained by two different processes, the actual one at Vascutek and the one by numerical simulation performed by Predisurge company.

ELIGIBILITY:
Inclusion Criteria:

- abdominal aortic aneurysms suitable for treatment using Fenestrated AnacondaTM (Vascutek) device

Exclusion Criteria:

* failure to generate an adequate FE model of patient arteries (no preoperative multidetector contrast-enhanced CT-scan available, preoperative CT-scan slice thickness greater than 1mm, preoperative CT-scan with artifacts)
* stent-graft setup implanted during the surgical procedure has been modified compared to preoperative planning
* patient refusing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have an abdominal aortic aneurysms treated by fenestrated endovascular anacondaTM of society Vascutek will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-22 (Actual)

PRIMARY OUTCOMES:
Vascutek in vitro validation test and the numerical simulation | Months: 18
  To compare Vascutek in vitro validation test and the numerical simulation (Predisurge). The proportion of fenestrations is less or equal to 2.5mm will be calculated.

SECONDARY OUTCOMES:
initial and final stent-graft designs obtained from Vascutek | Months: 18
  To study differences between initial and final stent-graft designs obtained from Vascutek process, the differences between L2 and L1 and C2 to C1 will be computed:
  L = for each fenestration, the longitudinal distance between centre of fenestration and top of fabric C = for each fenestration, circumferential angular distance between O° line and center of fenestration
  Current Vascutek protocol:
  * Initial custom Stent Graft design, right before in vitro testing = L1 and C1
  * Final custom Stent Graft design, after in vitro tests and subsequent design changes =L2 and C2
stent-graft designs obtained from simulation of deployment | Months: 18
  To study differences between stent-graft designs obtained from simulation of deployment in the polymer model and from simulation of deployment in the patient, the differences between L4 and L3 and C4 to C3 will be computed:
  L = for each fenestration, the longitudinal distance between centre of fenestration and top of fabric C = for each fenestration, circumferential angular distance between O° line and center of fenestration
  Simulation for fenestration positioning:
  * Initial custom Stent Graft design, right before in vitro testing = L3 and C3
  * Final custom Stent Graft design, after in vitro tests and subsequent design changes =L4 and C4

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand CHAVENT, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (9):
- Wilhelminen hospital, Vienna, Austria
- France (4):
  - CHU Bordeaux, Bordeaux
  - CHU Lyon, Lyon
  - Hôpitaux privés de Metz, Metz
  - Chu Saint-Etienne, Saint-Etienne
- University Hospital, Campus Benjamin Franklin, Berlin, Germany
- Netherlands (2):
  - Rijnstate Hospital, Arnhem
  - University Hospital Utrecht, Utrecht
- Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No